CLINICAL TRIAL: NCT03012087
Title: Using m-Health Tools to Reduce the Misuse of Opioid Pain Relievers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MyHealthyChoices
Record Dates: First submitted 2016-12-13; First posted 2017-01-06 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Prescription Drug Abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Risk Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): MyHealthyChoices
  Interventions: Behavioral: MyHealthyChoices
- Control Group (Placebo Comparator): Health Risk Assessment
  Interventions: Other: Health Risk Assessment

INTERVENTIONS:
Behavioral: MyHealthyChoices — My Healthy Choices explains what opioid pain medications are, assesses and explains the patient's risk factors related to taking opioids, assesses patient preferences about pain medications, and produces a tailored patient report based on the answers. The patient is encouraged to show the report to the treating ED clinician so they can discuss medication options for treating the patient's pain. Following discharge from the ED, intervention group participants discharged with a prescription pain reliever receive messages about safe medication use, storage, and disposal and access to an educational web portal that contains more information on prescription pain medications and safety.
  Arms: Intervention Group
Other: Health Risk Assessment — The WellSource health risk assessment content focuses on general health promotion, and the participant's overall health and wellness. A summary report based on the participants' answers is sent to their email address.
  Arms: Control Group

SUMMARY:
The aim of this study is to pilot test a web-based, patient-centered educational program that encourages the patient to have an informed discussion about pain medication options with their emergency department (ED) provider.

DETAILED DESCRIPTION:
This multi-site, randomized trial will evaluate an m-health program designed to aid the patient in making an informed decision about their pain treatment. Patients reporting to the ED with an injury-related chief complaint who agree to participate are randomized to receive the intervention program, My Healthy Choices, or an attention-matched control. My Healthy Choices pairs tailored education with a patient decision aid to describe what opioid and non-opioid pain medications are, assess the patient's risk factors for opioid-related adverse effects, and produce a tailored report that patients are encouraged to share with their doctor. Data are collected through surveys at three time points during the ED encounter (baseline, immediately after the intervention, and just before discharge), and at a 6-week follow-up survey. The primary outcomes are whether the patient prefers an opioid pain reliever (OPR) and whether the patient takes an OPR. The investigators hope this program will facilitate patient-provider communication, as well as reduce the number of prescriptions written for OPRs and thus the number of patients exposed to prescription opioids and the associated risks of addiction and overdose.

ELIGIBILITY:
Inclusion Criteria:

1. ED visit for an injury- or pain-related chief complaint
2. 18 years of age or older
3. speak English
4. has a smart phone or email address that is used on a regular basis
5. no previous medical care for the current complaint
6. triage pain score between 7-10

Exclusion Criteria:

* allergy to pain medications
* have used a prescription pain medication for more than two days in the past month
* report renal problems or a history of dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in Self-Reported Preference for Opioid Pain Reliever | Baseline and Immediate Post-test
  Assessed via questionnaire on a scale of 0-10.

SECONDARY OUTCOMES:
Change in Knowledge about Prescription Pain Medication Side Effects and Safe Practices for Taking, Storing and Disposing Prescription Pain Medications | Baseline and 6 weeks
  Assessed with a 25-item questionnaire. Knowledge items will be scored correct or incorrect and summed to generate a total knowledge score.
Self-Reported Prescription Drug Storage and Disposal Behaviors | 6 weeks
  Assessed via 5 items on a questionnaire. Behaviors will be scored correct or incorrect and tabulated across study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea C Gielen, ScD ScM, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - Johns Hopkins Hospital Emergency Department, Baltimore, Maryland
  - West Virginia University Emergency Department, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Omaki E, Castillo R, Eden K, Davis S, McDonald E, Murtaza U, Gielen A; My Healthy Choices Decision Aid Study Team. Using m-health tools to reduce the misuse of opioid pain relievers. Inj Prev. 2019 Aug;25(4):334-339. doi: 10.1136/injuryprev-2017-042319. Epub 2017 Apr 6. PMID 28385954